CLINICAL TRIAL: NCT04199637
Title: The Anxiety and Resisting Behavior Evaluation of Therapeutic Video Games for Pre-school Children With Acute Lymphoblastic Leukemia: Randomized Controlled Trial
Brief Title: Evaluation of Therapeutic Video Games for Pre-school Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, I-Ching Hou, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201705014RINC
Record Dates: First submitted 2019-11-19; First posted 2019-12-16 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Childhood Lymphoblastic Lymphoma
Keywords: Acute lymphoblastic leukemia; Therapeutic Video games; Childhood cancer; Preschoolers; Anxiety; Resisting behavior
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group is provided therapeutic video games
  Interventions: Other: TVG
- Control group (No Intervention): Control group is provided regular care

INTERVENTIONS:
Other: TVG — Therapeutic video game
  Arms: Experimental group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of therapeutic video game.

DETAILED DESCRIPTION:
Children cancer was the third-ranked causes of children's death. During the long treatment courses, children are always forced to accept lots of drug therapy and invasive procedures without understanding the medical purpose. Due to the immature cognition, always lead to anxiety in childhood cancer patients. Our team developed a mobile technology platform based therapeutic video game (TVG) for preschoolers with acute lymphoblastic leukemia (ALL) in early 2018. Then three clinical experts were invited to validate TVG and had high appropriateness consensus. Then the pilot study was conducted in one medical center in Taipei and 10 preschoolers with ALL had been randomly signed in two groups-5 to intervention group (6 weeks game intervention) and 5 to control group (regular care). The preliminary results showed that crying scale and resisting behavior were no significance between two groups in the initial period (p=.663), but the intervention group showed lower crying grades and less resisting behavior than the control group in the final period (p=.028). The limitation of this pilot research was small sample size and short intervention time. Therefore, the purpose of this study is to increase the sample size and intervention time to evaluate the effectiveness of our TVG.

Methods: A total of 68 fresh ALL preschool children will be randomized divided equally into intervention group and control group. Only intervention group

ELIGIBILITY:
Inclusion Criteria:

* ALL

Exclusion Criteria:

* non TPOG therapy
* without Port-A
* under PBST treatment
* ALL recurrent
* mental retardation

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The change of face pain rating scale | The continuous 8 weeks after recruiting
  Face pain rating scale(0 means for no hurt; 10 means for hurts worst) is measured by participants' family after receiving invasive therapies for continuous 8 weeks after recruiting.

CONTACTS AND LOCATIONS:
Overall Officials: IChing Hou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang DJ, Lu MY, Chen CW, Liu PC, Hou IC. Development of a Therapeutic Video Game With the MDA Framework to Decrease Anxiety in Preschool-Aged Children With Acute Lymphoblastic Leukemia: Mixed Methods Approach. JMIR Serious Games. 2022 Aug 22;10(3):e37079. doi: 10.2196/37079. PMID 35994340